CLINICAL TRIAL: NCT03044821
Title: Open Fetal Myelomeningocele Repair With Maternal BMI Between 35.0 And 40.0
Brief Title: Open Myelomeningocele Repair With High Maternal BMI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We now offer the repair as standard of care up to BMI of 40.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Michael Belfort, Professor and Chairman, Department of Obstetrics and Gynecology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-38734
Record Dates: First submitted 2016-05-24; First posted 2017-02-07 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Neural Tube Defect
Keywords: Neural Tube Defect
MeSH Terms: conditions — Neural Tube Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-Uterus Fetal Repair (Experimental): Single arm study. All patients will receive the open-uterus fetal repair.
  Interventions: Procedure: Open-Uterus Fetal Repair

INTERVENTIONS:
Procedure: Open-Uterus Fetal Repair — Single arm study. All patients will receive the open-uterus fetal repair.

SUMMARY:
Spina bifida is a neurological abnormality characterized by an opening in the skin and exposure of the spinal cord on the back of the baby at the time of birth. The complete closure and separation of the spinal cord from the skin occurs in the first month of pregnancy.

This form of spina bifida is associated with leg weakness, sensation loss, and bowel and bladder incontinence. The majority of patients (>80%) also develop increased fluid in the brain, called hydrocephalus, and require additional surgery to treat this problem. Standard treatment of myelomeningocele (MMC) involves closing the opening in the back within the first 3 days of life. The surgery releases the spinal cord from the skin and brings the skin edges together to prevent infection and injury to the exposed nerves. Of note, this type of surgery does not improve function.

The investigators want to study the open in-utero fetal surgery technique in patients who are candidates for the standard open fetal repair technique but have a pre-pregnancy BMI of 35.0-40.0. The latter is a reason for exclusion for open fetal repair in most centers in the United States.

DETAILED DESCRIPTION:
The research will be conducted at the following location(s):

Baylor College of Medicine and Texas Children's Hospital- Women's Pavilion.

About 15 subjects will be enrolled in this study. In order to be eligible for this study, the participant must meet the established criteria for open fetal MMC surgery but also have a BMI of 35.0-40.0.

PREOPERATIVE AND INTRAOPERATIVE CONCOMITANT MEDICATIONS:

The participant will receive two doses of 12 mg betamethasone, 24 hours apart, for fetal lung maturation if the gestational age is greater than 23 weeks. The participant will also receive the prophylactic tocolysis (medications to prevent preterm contractions) indomethacin 50 mg prior to surgery, then 25-50 mg every six to eight hours for 24-48 hours following the surgery, longer if clinically indicated. Magnesium sulfate may also be used intraoperatively - 6 gram IV loading dose followed by a 2 gram/hour continuous infusion for 24 - 72 hours. In addition, if medically indicated, nifedipine (10mg orally) or terbutaline (0.25mg subcuticularly) may be substituted for the indomethacin or magnesium sulfate based on condition and medical judgment. Prophylactic antibiotics will also be administered to the participant prior to the procedure using cefazolin, azithromycin, and/or metronidazole, or if medical history contraindicates the use of cefazolin, clindamycin,azithromycin, and gentamicin will be administered. A solution of nafcillin and lactated ringers will be injected into the amniotic cavity at the conclusion of the procedure. Additional medications, including therapeutic antibiotics, may be used as part of standard of care by the medical team.

MATERNAL-FETAL ANESTHESIA:

The participant will have a lumbar epidural catheter placed prior to surgery for postoperative analgesia. The procedure will be performed under general anesthesia following a rapid sequence intubation with propofol and succinylcholine. Anesthesia will be maintained with 2-3 times MAC (Minimal anesthetic concentration) of volatile anesthetic agent. This high concentration of anesthetic agent provides adequate uterine relaxation during surgery. After the defect has been repaired and once closure of the skin incisions begins, local anesthetic will be administered through the epidural catheter and the participant will be started on a continuous epidural infusion of local anesthetic and opioid combination. The participant will receive this medication via an epidural pump for approximately 3-4 days following surgery. The epidural pump has the capability of the patient self-administering intermittent boluses of medication on top of the continuous infusion rate if the participant becomes uncomfortable in the post-operative period.

The fetus will receive an intramuscular injection of opioid (fentanyl 5-10 mcg/kg), anticholinergic (atropine 20 mcg/kg), and muscle relaxant (vecuronium 0.3 mg/kg) into the buttock or extremity using a 22G needle that is passed through the port in order to provide muscle relaxation, sedation, and analgesia. The drug dosages are adjusted to the estimated fetal weight. The fetus will receive the injection prior to starting the CO2 gas insufflation into the uterus and will continue to receive the combo injection approximately every 45 - 60 minutes throughout the remainder of the procedure as deemed necessary by the medical team.

Subsequent combo injections will be administered by passing the 22G needle through one of the uterine ports. General maternal anesthesia with anesthetic gases is known to provide fetal anesthesia. The combination injection will provide muscle relaxation and additional analgesia to the fetus. This combination of medications is routinely administered to fetuses during open fetal surgery and has been found to adequately sedate the fetus during fetal intervention procedures.

SURGICAL REPAIR:

The investigators will either make a lower transverse incision (also called the 'bikini cut') or a midline vertical incision to gain access to the uterus. The incision will be about the same size (about 8-10 inches) that is needed for a typical cesarean section procedure. Once the uterus is exposed an ultrasound will be performed to determine the position of the fetus for the surgery and cardiac function will be monitored. If necessary, the fetus will be gently repositioned from outside the uterus so that the fetal back is facing upwards. Ultrasound will be used to help the surgical team determine the position of the fetus at all times.

The fetus will receive an anesthesia injection into the buttock or thigh prior to the start of the repair. The anesthesia injection is a combination of medications that block pain and help relax the muscles. In addition, maternal anesthesia is also known to provide anesthesia to the fetus.

When the defect is clearly identified, the spinal cord will be released from its attachments to the skin. The skin edges will be sewn together using an absorbable suture and repair technique similar to the standard technique in women with BMI<35.0. Sometimes it might be better to use one type or style of suture (surgical thread) during the surgery. While this can be generally the same from one patient to the next, it may be in the participating mother's or fetus's best interest to change the suture or suture technique to adapt to the surgery being performed.

All pre- and post-operative care and all follow-up visits are the same as with any open procedure and are considered standard of care; therefore, the participant will not be responsible for any costs related to this research study other than the normal co-pays or deductibles. Following the participant's discharge from the hospital, the participant will need to stay within a 30-minute drive of Texas Children's Hospital Pavilion for Women to allow for medical care after the operation. The participant will be responsible for any accommodation costs in Houston.

POSTOPERATIVE FOLLOW-UP:

The investigators will collect clinical information from the participant's medical chart during standard clinical care. In addition, the investigators will collect clinical information about the participating child until he/she turns 5 years old. The following information will be collected from clinical records of the participating mom and child : 1. Demographics (age, parity, height, weight, BMI, use of drugs and alcohol, smoking, clinical disease, medications, medical history); 2. Prenatal data (gestational age, ultrasound and MRI findings, results of amniocentesis, vital signs) 3. Fetal intervention (surgery information, gestational age, complications, post-procedure follow-up including ultrasound); 4. Intra-partum data (ultrasound and MRI findings, gestational age at delivery, type of labor, mode of delivery, indications and complications, status of port sites if cesarean delivery); 5. Immediate neonatal period data (birth weight, Apgar scores, physical exam findings, hydrocephalus assessment, repair site condition, imaging, need for surgery or shunt placement, imaging results); 6. Long-term follow-up every 3-4 months in the first year, Year 1, Year 2, Year 3, Year 4, and Year 5 (physical exam findings, imaging results, and hydrocephalus assessment).

Like all children with spina bifida, the participating child will be taken care of by the pediatric neurosurgery service after birth. Follow-up visits occur in the Spina Bifida Clinic at Texas Children's Hospital. All follow up visits are considered standard of care and will occur as follows:

After the baby is born, and before they leave the hospital, they will have a physical exam, an assessment of hydrocephalus, urinary and orthopedic evaluations, and imaging of their brain.

In the first year, the child will have a visit every 3-4 months where a physical exam and urinary and orthopedic evaluations will be done. Year 1 and Year 2 visits will include: a physical exam, developmental assessment, urinary and orthopedic evaluations, and an assessment for hydrocephalus. The Year 1 visit will also include imaging of the child's brain and spine (this may be repeated if needed at any point).

At Year 3 and Year 4, a physical exam and urinary and orthopedic evaluations will be done.

Year 5 is the end of participation in this study. This visit will include: a physical exam, developmental assessment, assessment for hydrocephalus and imaging of the child's spine and head.

After Year 5, there will be routine annual follow up visits. If the participant moves away from Texas, the investigators will attempt to follow up with a review of the mom and child medical records The participant will be asked to sign a medical record release, every year if needed, to allow this to occur. The participant may be contacted by study staff regarding any changes to the study and asked to sign a new informed consent form. The participant may be contacted by phone by study staff about the medical release form or changes to the study.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women - maternal age 18 years or older and capable of consenting for their own participation in this study.
2. Singleton pregnancy
3. MMC with the upper boundary located between T1 and S1
4. Evidence of hindbrain herniation (confirmed on MRI to have an Arnold-Chiari type II malformation).
5. Absence of chromosomal abnormalities and associated anomalies
6. Gestational age at the time of the procedure will be between 19 0/7 weeks and 25 6/7 weeks
7. Normal karyotype and/or normal chromosomal microarray (CMA) by invasive testing (amniocentesis or CVS). If there is a balanced translocation with normal MCA with no other anomalies the candidate can be included. Patients declining invasive testing will be excluded.
8. Family has considered and declined the option of termination of the pregnancy at less than 24 weeks.
9. Family meets psychosocial criteria (sufficient social support, ability to understand requirements of the study).
10. Parental/guardian permission (informed consent) for follow up of child after birth.

Exclusion Criteria:

1. Fetal anomaly unrelated to MMC.
2. Severe kyphosis.
3. Increased risk for preterm labor including short cervical length (<1.5 cm), history of incompetent cervix with or without cerclage, and previous preterm birth.
4. Placental abnormalities (previa, abruption, accreta) known at time of enrollment
5. A pre-pregnancy body-mass index ≥35
6. Contraindications to surgery including previous hysterotomy (whether from a previous classical cesarean, uterine anomaly such as an arcuate or bicornuate uterus, major myomectomy resection, or previous fetal surgery) in active uterine segment.
7. Technical limitations precluding fetoscopic surgery, such as uterine fibroids, fetal membrane separation, uterine anomalies incompatible with fetoscopy.
8. Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy.
9. Maternal HIV, Hepatitis-B, Hepatitis-C status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis status is unknown, the patient must be tested and found to have negative results before enrollment.
10. Maternal medical condition that is a contraindication to surgery or anesthesia.
11. Low amniotic fluid volume (Amniotic Fluid Index less than 6cm) if deemed to be due to fetal anomaly, poor placental perfusion or function, or membrane rupture. Low amniotic fluid volume that responds to maternal hydration is not an exclusion criterion.
12. Patient does not have a support person (ie. Spouse, partner, mother) available to support the patient for the duration of the pregnancy.
13. Inability to comply with the travel and follow-up requirements of the trial.
14. Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy
15. Patient scores as severely depressed on the BDI-II questionnaire; a score of 29 or above.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Complications associated with obesity during Surgery. | At the time of fetal repair surgery.
  Determine if there is an increased risk for mothers with a BMI of 35-40 during an open in-utero surgical repair for myelomeningocele.
Complications associated with obesity during pregnancy. | During the post-surgical course of pregnancy.
  Determine if there is an increased risk for mothers with a BMI of 35-40 after having undergone an open in-utero surgical repair for myelomeningocele.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Belfort, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States